CLINICAL TRIAL: NCT05980117
Title: Comparison of Remimazolam vs. Midazolam for Sedation During Cataract Surgery
Brief Title: Remimazolam for Cataract Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhuang T. Fang, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-001570
Record Dates: First submitted 2023-06-21; First posted 2023-08-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cataract Surgery; Cognitive Impairment
Keywords: Midazolam; Remimazolam; Outcomes
MeSH Terms: conditions — Cognitive Dysfunction | interventions — remimazolam; Midazolam

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the intervention group receiving Remimazolam or to the control group receiving Midazolam.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Patients assigned to the study group will receive Remimazolam.
  Interventions: Drug: Remimazolam
- Control (Active Comparator): Patients assigned to the control group will receive Midazolam.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam (1.0mg IV) titrated to modified observer's assessment of sedation score of 3 -4 during cataract surgery.
  Other Names: Byfavo
  Arms: Intervention
Drug: Midazolam — Midazolam (0.5-2mg IV) titrated to modified observer's assessment of sedation score of 3 - 4 during cataract surgery.
  Other Names: Versed
  Arms: Control

SUMMARY:
The goal of this study is to assess any post operative cognitive changes following benzodiazepine administration during cataract surgery. The investigators will compare effects of Midazolam vs. Remimazolam on cognition at the time of discharge from the post operative care unit and the next day following surgery.

Cognitive changes will be assessed by administration of Montreal Cognitive Assessment (MoCA).

Participants will:

1. Complete MoCA testing prior to surgery
2. Randomize in either Midazolam or study drug Remimazolam
3. Complete MoCA testing after surgery at the time of discharge in the post anesthesia care unit and the next day of surgery at the time of post operative surgical visit.
4. Complete Patient Satisfaction Survey at the time of discharge from the Post Anesthesia Care Unit (PACU)

DETAILED DESCRIPTION:
Cataract surgery (clouded natural lens of eye removed and clear artificial lens implanted) is the most common eye surgery performed in elderly patients. Although cataract surgery is a minor surgery, many patients are anxious and therefore benzodiazepine such as midazolam is administered during surgery to allay a patient's anxiety.

The purpose of this study is to look at any difference in postoperative cognitive changes as well as recovery times in the PACU following administration of midazolam or remimazolam.

Patients will be asked to participate in a clinical trial where they will be randomly assigned to midazolam or remimazolam group. Cognitive changes will be assessed by administration of MoCA test. MoCA test is a validated, objective short (about 10-15 minutes) screening tool for detection of mild neurocognitive dysfunction. Given the short half life of remimazolam, investigators hypothesize that any cognitive changes will be less with remimazolam compared to midazolam.

Patients will be asked to complete MoCA prior to surgery, in the recovery room following surgery, and the next day during their post-operative clinic visit. In addition, patients will be asked to rate their satisfaction of their anesthetic during their surgery.

The participant will be in this research study from the day of surgery until the first post-operative visit, the following day.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age > 65 years undergoing first eye cataract surgery under local topical anesthesia at the University of California, Los Angeles (UCLA).
2. Both male and female patients
3. American Society of Anesthesiologists Class 2, 3, and 4.

Exclusion Criteria:

1. Patients who are unable to consent for the study
2. Patients who are unable to cooperate with the cognitive assessment such as patients with significant visual, auditory, language or other impairment.
3. Patients who are unable to understand simple English commands.
4. Patients who do not wish to have benzodiazepine medication during surgery
5. Patients with a history of severe hypersensitivity reaction to dextran 40 or products containing dextran 40.
6. Patients with chronic pain on opiates.
7. Patients with a history of drug, alcohol abuse/dependence.
8. Patients with BMI > 40.
9. Patients with obstructive sleep apnea (moderate to severe).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in MoCA score following surgery in the PACU and post operative day 1. | Immediately following surgery in the PACU and post operative day 1.
  Montreal Cognitive Assessment (MoCA) test. A numerical scale is used for scoring. 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment
Change in MoCA Scores in PACU and the next day between midazolam and remimazolam group. | Immediately following surgery in the PACU, and post operative day 1.
  Montreal Cognitive Assessment (MoCA) test. The following ranges may be used to grade severity: A numerical scale is used for scoring. 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment.
Length of postoperative stay | Postop day 0 (day of surgery) until discharge from the hospital, usually on postop day 1 (an average of 1 day).
  Duration from the time of admission to readiness for discharge from the PACU. The following ranges may be used to grade severity:

SECONDARY OUTCOMES:
Surgeon Satisfaction | Intraoperatively to postoperatively in the ICU, and expected average of 1 hour.
  Surgeon satisfaction score will be assessed post-surgery as measured by a 5-point scale with 1 = Strongly Disagree , 2 = Disagree , 3 = Neither Agree nor Disagree, 4 = Agree, 5 = Strongly Agree.
Patient Satisfaction | Day of surgery
  Patient satisfaction score will be assessed at the time of discharge by a 5 point scale with 1 = Disagree Strongly , 2 = Disagree Somewhat , 3 = Neither Agree or Disagree, 4 = Agree Somewhat, 5 = Agree Strongly.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Fang, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rabinowitz LE, Lamper L, Tendler JM, Schlesinger JM, Vera N. Preventing Adverse Events in Cataract Surgery. Anesth Analg. 2018 Oct;127(4):e66. doi: 10.1213/ANE.0000000000003655. No abstract available. PMID 30059403
- [Background] Chung F, Lavelle PA, McDonald S, Chung A, McDonald NJ. Cognitive impairment after neuroleptanalgesia in cataract surgery. Anesth Analg. 1989 May;68(5):614-8. PMID 2719292
- [Background] Evered LA, Silbert BS, Scott DA, Maruff P, Ames D, Choong PF. Preexisting cognitive impairment and mild cognitive impairment in subjects presenting for total hip joint replacement. Anesthesiology. 2011 Jun;114(6):1297-304. doi: 10.1097/ALN.0b013e31821b1aab. PMID 21502855
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Tan Y, Ouyang W, Tang Y, Fang N, Fang C, Quan C. Effect of remimazolam tosilate on early cognitive function in elderly patients undergoing upper gastrointestinal endoscopy. J Gastroenterol Hepatol. 2022 Mar;37(3):576-583. doi: 10.1111/jgh.15761. Epub 2022 Jan 3. PMID 34907594